CLINICAL TRIAL: NCT01553682
Title: Reducing Alcohol-Related HIV Risk in African American Females
Brief Title: Project N-Liten- HIV Prevention for African American Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Ralph J. DiClemente, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00048502; 5R01AA018096 (NIH)
Record Dates: First submitted 2012-03-05; First posted 2012-03-14 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: Sexually Transmitted Diseases
Keywords: HIV; STDs; African American Females; Alcohol
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Enhanced Standard-Of-Care (No Intervention): Participants will watch a video about how to prevent STIs and HIV, then do question and answer session. This group will be last 1 hour. It will be led by one African American health educator, and have about 4-8 other young women participants. Participants will be asked to rate the workshop anonymously.
- Horizons+General Health Promotion (GHP) (Active Comparator): Participants will attend the Horizons HIV Prevention Program with an extra workshop on nutrition health promotion. Participants will attend a total of two (2) 5-hour workshops over 2 consecutive Saturdays. They will be led by African American health educators, and have about 8-12 other young women participants. The workshops will discuss gender and ethnic pride, self-esteem, good role models, and how to reduce risky sexual behavior. The nutrition health promotion workshop will give ideas on healthy nutrition and exercise. Participants will be asked to rate the workshop anonymously.
  Interventions: Behavioral: Horizons+General Health Promotion (GHP)
- Horizons+Motivational Enhancement Therapy (GMET) (Experimental): Participants will attend the Horizons Plus HIV Prevention Program. Participants will attend a total of two (2) 5-hour workshops over 2 consecutive Saturdays. They will be led by African American health educators, and have about 8-12 other young women participants. The workshops will discuss gender and ethnic pride, self-esteem, good role models, and how to reduce risky sexual behavior. Participants will be asked to rate the workshop anonymously.
  Interventions: Behavioral: Horizons+Motivational Enhancement Therapy (GMET)

INTERVENTIONS:
Behavioral: Horizons+General Health Promotion (GHP) — Participants will attend the Horizons HIV Prevention Program with an extra workshop on nutrition health promotion. Participants will attend a total of two (2) 5-hour workshops over 2 consecutive Saturdays. They will be led by African American health educators, and have about 8-12 other young women participants. The workshops will discuss gender and ethnic pride, self-esteem, good role models, and how to reduce risky sexual behavior. The nutrition health promotion workshop will give ideas on healthy nutrition and exercise. Participants will be asked to rate the workshop anonymously.
  Arms: Horizons+General Health Promotion (GHP)
Behavioral: Horizons+Motivational Enhancement Therapy (GMET) — Participants will attend the Horizons Plus HIV Prevention Program. Participants will attend a total of two (2) 5-hour workshops over 2 consecutive Saturdays. They will be led by African American health educators, and have about 8-12 other young women participants. The workshops will discuss gender and ethnic pride, self-esteem, good role models, and how to reduce risky sexual behavior. Participants will be asked to rate the workshop anonymously.
  Arms: Horizons+Motivational Enhancement Therapy (GMET)

SUMMARY:
Young African-American women who report a higher frequency of alcohol use have particularly higher rates of sexually transmitted diseases (STDs) and human immunodeficiency virus (HIV) sex behaviors. Unfortunately, there are no evidence-based HIV interventions designed to be gender- and culturally-appropriate for this population. To address this, the investigators propose to add to the CDC-defined evidence-based intervention (DEBI), Horizons, a new intervention form, Group Motivational Enhancement Therapy (GMET), which has shown promise in reducing alcohol use and alcohol-related HIV risk-taking. To test how effective the combined Horizons+GMET alcohol-specific portion is, it will be evaluated with a time equivalent Horizons+attention control general health promotion (GHP) portion focusing on nutrition health promotion, and to an enhanced standard-of-care program. In this study, 600 young African American women, 18-24 years of age, who report 3 or more occasions where they drank alcohol in the past 90 days will be recruited to complete a four-part baseline assessment consisting of: 1. an audio computer assisted self interview (ACASI), 2. videotaped communication role plays to objectively measure communication skill ability (subsample), 3. provide a vaginal specimen to test for STDs and 4. Provide a urine pregnancy screen. After participants complete their baseline assessment, they will be randomly assigned to one of three conditions: 1. Horizons+GMET alcohol-specific condition, 2. a time-equivalent Horizons+GHP condition, or 3. an enhanced standard-of-care control condition. The GMET alcohol-specific component has shown to be effective in influencing several alcohol-specific concepts (attitudes, norms, self-efficacy) and reducing sexual risk-taking among culturally-diverse high-risk youth. The GMET alcohol-specific module was designed to increase woman's awareness of the unfavorable effects of alcohol on themselves, their sexual decision-making, and their male partner and teaches women strategies to reduce the possibility of engaging in sex under the influence of alcohol. In addition, the GMET alcohol-specific module provides skills training needed to effectively talk about sexual intentions to use condoms and/or refuse risky sex when they or their male sex partner has been using alcohol. After completing one of the three conditions, participants will complete a brief ACASI posttest to evaluate immediate changes in hypothesized social and psychological mediators of safer sex and alcohol use. Participants will also return to complete follow-up assessments at 3, 6, 9, and 12-months after their intervention. If the Horizons+GMET intervention is observed to be effective, investigators will work closely with the CDC DEBI program to help distribute the intervention to public health agencies and community based organizations (CBOs).

ELIGIBILITY:
Inclusion Criteria:

* To be eligible, participants must be:

  * African American women;
  * 18-24 years of age, inclusive at time of enrollment;
  * unmarried;
  * report having at least one episode of unprotected vaginal or anal sex in the past 90 days;
  * report ≥ 3 alcohol drinking episodes in the past 90 days;
  * not pregnant; and
  * provide written informed consent.

Exclusion Criteria:

* Those with:

  * the presence of active psychosis reflected by the participant's status during the baseline assessment, and/or
  * an acute or chronic illness that could preclude participation for the duration of the program and follow-up will be excluded.

Ages: 18 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 560 (Actual)
Dates: Start 2011-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incident STD infection confirmed by laboratory PRC testing over a 12-month follow-up. | 12 months post-randomization
  Incident STD infection confirmed by laboratory PRC testing.

SECONDARY OUTCOMES:
Proportion of condom-protected vaginal or anal sex acts over a 12-month follow-up. | 12 months post-randomization
  Assessed by ACASI

CONTACTS AND LOCATIONS:
Overall Officials: Ralph J DiClemente, PhD, Principal Investigator — Emory University; Jennifer L. Monahan, PhD, Principal Investigator — University of Georgia
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] DiClemente RJ, Rosenbaum JE, Rose ES, Sales JM, Brown JL, Renfro TL, Bradley ELP, Davis TL, Capasso A, Wingood GM, Liu Y, West SG, Hardin JW, Bryan AD, Feldstein Ewing SW. Horizons and Group Motivational Enhancement Therapy: HIV Prevention for Alcohol-Using Young Black Women, a Randomized Experiment. Am J Prev Med. 2021 May;60(5):629-638. doi: 10.1016/j.amepre.2020.11.014. Epub 2021 Mar 5. PMID 33678517